CLINICAL TRIAL: NCT02292160
Title: Does the National Health Insurance Card Allow us to Predict Antibiotic Resistance? Pilot Study to Guide Probabilistic Antibiotic Regimens of Community-acquired Urinary Tract Infections
Brief Title: Does the National Health Insurance Card Allow us to Predict Antibiotic Resistance?
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/186/HP
Record Dates: First submitted 2014-10-20; First posted 2014-11-17 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Urinary Tract Infection Empiric Antibiotic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective is to determine if data from the National Insurance Health card (giving antibiotics and hospitalizations in the past 18 months) allow to predict the individual risk of antibiotic resistance and to identify population groups for which probabilistic antibiotics regimen of urinary tract infection could be simplified

ELIGIBILITY:
Inclusion Criteria:

* national health insurance card available
* community acquired urinary tract infection

Exclusion Criteria:

* incapacity to accept an inform consent
* hospitalized acquired urinary tract infection
* national health insurance card non available

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with an community-acquired urinary tract infection
Sampling Method: Probability Sample
Enrollment: 1128 (Actual)
Dates: Start 2015-09; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Frequency of antibiotic resistant organisms | One year
  Frequency of antibiotic resistant organisms in patient with urinary infection

CONTACTS AND LOCATIONS:
Overall Officials: Francois CARON, Pr, Principal Investigator — UH Rouen
Locations (2):
- France (2):
  - Lbmr de Normandie, Elbeuf
  - Rouen University Hospital, Rouen

REFERENCES:
- [Derived] Vautrin N, Dahyot S, Leoz M, Caron F, Grand M, Feldmann A, Gravey F, Legris S, Ribet D, Alexandre K, Pestel-Caron M. Are Escherichia coli causing recurrent cystitis just ordinary uropathogenic E. coli (UPEC) strains? Virulence. 2025 Dec;16(1):2444689. doi: 10.1080/21505594.2024.2444689. Epub 2024 Dec 26. PMID 39726097
- [Derived] Alexandre K, Reveillon-Istin M, Fabre R, Delbos V, Etienne M, Pestel-Caron M, Dahyot S, Caron F. Temocillin against Enterobacteriaceae isolates from community-acquired urinary tract infections: low rate of resistance and good accuracy of routine susceptibility testing methods. J Antimicrob Chemother. 2018 Jul 1;73(7):1848-1853. doi: 10.1093/jac/dky101. PMID 29635629